CLINICAL TRIAL: NCT06927141
Title: Effect of Flexible Catheter Materials on Catheter Angle, Dwell Time, Thrombosis and Interstitial Oedema
Brief Title: Effect of Flexible Catheter Materials on Catheter Angle and Blood Vessel Irritation
Acronym: FLEXIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffith University (Other)
Collaborators: Queensland University of Technology (Other); University of Galway (Other); Poitiers University Hospital (Other); Terumo Corporation (Industry); Queensland Health (Other Government)
Responsible Party: Principal Investigator, Andrew Bulmer, Professor, Griffith University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/150
Record Dates: First submitted 2025-03-27; First posted 2025-04-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Intravenous Catheterization; Oedema; Thrombosis
Keywords: Catheter Angle; Interstitial Oedema; Peripheral Intravenous Catheter; Catheter Materials; Indwell; Cannulation; FLEXIT; Vascular Access Device
MeSH Terms: conditions — Edema; Thrombosis | interventions — Catheterization

STUDY DESIGN:
Intervention Model Description: Two catheters are being compared simultaneously using a bilateral cannulation model. Participants will be randomised for which catheter will be inserted into either arm, but all participants will be cannulated with both catheters. The randomisation algorithm will be designed to ensure that left- and right-hand dominant participants are distributed evenly across treatment arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left More Flexible Right Less Flexible (Experimental): Participants in this arm will have a more flexible catheter placed in their left arm.
  Interventions: Device: Bilateral Peripheral Intravenous Catheterisation
- Left Less Flexible Right More Flexible (Experimental): Participants in this arm will have a less flexible catheter placed in their left arm.
  Interventions: Device: Bilateral Peripheral Intravenous Catheterisation

INTERVENTIONS:
Device: Bilateral Peripheral Intravenous Catheterisation — Participants will have peripheral intravenous catheters inserted. Each participant will receive two different catheters (less flexible = 20 gauge ICUMedical SuperCath5 SP120-20-31T; more flexible = 20 gauge Becton Dickinson Insyte Autoguard Blood Control 381034), with the treatment arm (more flexible) being randomly assigned.
  Other Names: Cannulation

SUMMARY:
Peripheral intravenous catheters (PIVCs; commonly known as "cannulas") are very small tubes made out of rubber-like materials which are inserted into patients' arms using a needle to allow easy access to veins. They are the most commonly-used medical devices in the world, with almost 10 million placed each year in Australia alone. Approximately 40% (almost 4 million) of these devices stop working (i.e. fail) prior to completion of therapy.

The main goal of this study is to learn if softer, more flexible PIVC tip materials reduce the angle of the catheter tip on the vein surface compared to less flexible materials. Reducing the angle of the tip is believed to reduce rubbing on the inner vein surface and causing irritation, extending the life of the catheter. Other goals of this study are to learn if softer materials affect: volume of oedema (i.e. fluid leakage around the vein); time until catheter failure; clot volume in the vein; changes in vein size in response to catheter insertion; adverse event rates (i.e. changes in rates of specific, reportable symptoms); and determining if certain catheters are better for some people than others. This study is recruiting participants of all genders aged 18 - 75 years old who:

* Are not pregnant
* Have a Body Mass Index (BMI) between 18.5 - 35 kg/m2
* Have a current Australian Medicare card
* Do not have a history of chronic/infectious disease or clotting disorders
* Do not have a history of recreational drug use or alcohol abuse within the past 2 years

Participants will:

* Spend two hours in the clinic for screening blood collection, medical questionnaire and ultrasound imaging of veins
* Have one more flexible catheter and one less flexible catheter placed in opposite arms (i.e. participants will have a total of two catheters placed) which will remain in place either (i) until they fail or (ii) for 72 hours, whichever is earlier
* Spend eight hours per day in the clinic on the day the catheters are placed and the two days following for observation and ultrasound imaging
* Spend four hours in the clinic on the third day following placement of the catheters for observation, ultrasound imaging and catheter removal
* Spend one hour in the clinic 24-96 hours after catheter removal for a follow-up assessment and questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-75 years.
* Not pregnant at time of recruitment and within 48 hrs of Day 1 procedures (self-reported)
* Normal haematology results as per reference range determined by the laboratory.
* Normal coagulation results as per reference range determined by the laboratory.
* Target cephalic veins readily cannulatable (i.e., > 2 mm)
* Able and willing to provide verbal and written consent
* Must be an Australian citizen with current Medicare card

Exclusion Criteria:

* History of pro coagulative state / condition (e.g., previous deep vein thrombosis)
* Currently on any anti-coagulant or platelet inhibitor medication. Use of NSAIDs and aspirin will be documented however are not exclusionary.
* Haemophilia or any current or history of bleeding disorder or tendency
* Presence or report of current blood borne disease/infection (e.g., hepatitis, HIV, leukemia, lymphoma)
* History of difficult vascular access
* Allergy or sensitivity to chlorhexidine gluconate, isopropyl alcohol, latex, or skin adhesives
* BMI < 18.5 kg/m2 or ≥ 35 kg/m2
* Positive results for the urine drug screen at screening or check-in (including opiates, methadone, cocaine, amphetamines)
* History or presence of alcoholism (self-reported) or drug abuse within the past 2 years
* A current or previous medical, physical, mental / cognitive disorder or anatomical conditions that, in the opinion of the chief or sub-investigator, would place the patient at risk, would make them unable to perform study procedures or has the potential to confound interpretation of the study results. (e.g., musculo-skeletal injury, chronic back pain)
* Employed by Terumo, Becton Dickinson, Teleflex Medical, ICUMedical or BBraun (conflict of interest)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Catheter Angle | Baseline (Day 1: morning)
  Measured against inferior border of vein using vascular ultrasound (in degrees)

SECONDARY OUTCOMES:
Volume of interstitial oedema | Morning visit (AM) after catheter insertion through to final interventional visit (up to 4 days)
  Measured using vascular ultrasound (in mm cubed/microliters)
Time to catheter failure | Morning visit (AM) after catheter insertion through to catheter removal and/or 72 hours post-insertion (whichever is earlier)
  Measured separately for each PIVC (in hours), including differences between catheters and survival analysis.
Thrombus volume in vein | Morning visit (AM) after catheter insertion through to catheter removal and/or 72 hours post-insertion (whichever is earlier)
  Measured using vascular ultrasound (in mm cubed/microliters)
Vein segment volume | Morning visit (AM) after catheter insertion through to catheter removal and/or 72 hours post-insertion (whichever is earlier)
  Measured by vascular ultrasound (in mm cubed/microliters)
Adverse Events | Morning visit (AM) after catheter insertion through to follow-up visit (up to 7 days)
  Identified by study team and/or nurses and reviewed by a medical practitioner (identified individually and aggregate of all adverse events; expressed as a count and percentage of catheters inserted).

OTHER OUTCOMES:
Multiple regression analysis | Screening until follow-up appointment (screening period indeterminate, follow-up appointment completed up to 7 days post-insertion)
  Determining independent predictors from demographic data (i.e. biological sex (M/F)) on outcome measures (catheter dwell/failure time, thrombus/vessel/oedema measrements, adverse events).
Multiple regression analysis | Screening until follow-up appointment (screening period indeterminate, follow-up appointment completed up to 7 days post-insertion)
  Determining independent predictors from demographic data (i.e. age (years)) on outcome measures (catheter dwell/failure time, thrombus/vessel/oedema measrements, adverse events).
Multiple regression analysis | Screening until follow-up appointment (screening period indeterminate, follow-up appointment completed up to 7 days post-insertion)
  Determining independent predictors from demographic (i.e. biological sex (M/F), age (years), height (cm), weight and height will be combined to report BMI in kg/m^2), family history of disease etc), haematologic (i.e. platelet, white/red blood cell counts [cells per microliter], clotting times [PT/APTT; sec], fibrinogen [mg/dL or g/L], DDimer [mg/L or ug/mL] etc and biochemical tests [liver [U/L] and kidney function tests mg/dL or umol/L], protein/s, petdides [ug/L or ng/mg protein], lipid profile (mmol/L), glucose (mg/dL or mmol/L) etc) on outcome measures (catheter dwell/failure time, thrombus/vessel/oedema measrements, adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Griffith University
Locations (1):
- Griffith University, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication in an international peer-reviewed journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning from first participant enrolment with no end date
Access Criteria: Only team members with direct participant interaction will have access to identifiable data. Other team members (e.g. statistician and computer scientists) will have access to de-identified data which will be limited only to that data which is necessary to complete their assigned role. The funder and general public will have access only to de-identified IPD that underlie results in the form of a published journal article. The funder and all members of the team will have access to the study protocol, SAP, ICF and CSR, but only team members listed on the Protocol have authority to influence/make changes to these documents.